CLINICAL TRIAL: NCT02726347
Title: Pneumococcal Post-Vaccination Titers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Flavia Hoyte, Principal Investigator, National Jewish Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-2953
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Smokers, Elderly, Asthma, COPD, Recurrent Infections
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Reinfection | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Smokers between the ages of 19-80 (Active Comparator): current smokers between the ages of 19 and 80
  Interventions: Biological: PPV-23
- elderly individuals (over age 50) (Active Comparator): elderly individuals, defined as subjects age 50 years or older, without a history of frequent infections, COPD, or asthma
  Interventions: Biological: PPV-23
- COPD subjects (Active Comparator): COPD subjects between the age of 19 and 80, without history of recurrent bacterial infections.
  Interventions: Biological: PPV-23
- Asthmatics subjects (Active Comparator): Asthmatics between the ages of 19 and 80
  Interventions: Biological: PPV-23
- Subjects with recurrent bacterial infections (Active Comparator): Individuals between the age of 19 and 80 who have a history of frequent bacterial infections and are being evaluated for humoral immunodeficiency
  Interventions: Biological: PPV-23

INTERVENTIONS:
Biological: PPV-23 — one hundred forty subjects will have pre-vaccination titers checked. All will be given vaccination as standard of care. Approximately 4 weeks later subjects will have post-vaccination titers checked for the same serotypes.
  Other Names: polysaccharide pneumococcal vaccine

SUMMARY:
The study is looking at the pneumonia vaccine and the immune system response to this vaccine. The information gathered from this study may be important for your doctor to take care of patients with smoking histories, immune deficiency, asthma, Chronic Obstructive Pulmonary Disease (COPD), or elderly patients. It is important that your immune system builds a strong defense to the vaccine so that you are better able to fight a bacterium that can cause pneumonia. Some disease prevent the immune system from building a strong defense and these patients will not benefit from the vaccine.

DETAILED DESCRIPTION:
One hundred forty subjects will have pre-vaccination titers checked for the 23 serotypes in the PPV-23 vaccine. They will then receive the vaccine. All subjects will be given the vaccination as standard of care. Approximately 4 weeks following immunization, the subjects will have post-vaccination titers checked to the same serotypes checked prior to vaccination.

ELIGIBILITY:
Inclusion Criteria:

Informed consent will be administered to individuals from 5 cohorts each with 28 subjects for a total of 140 subjects. The cohorts will be:

1. smokers between the ages of 19-80.
2. elderly individuals, defined as subjects age 50 years or older, without a history of frequent infections, COPD or asthma.
3. COPD subjects between the age of 19 and 80, without a history of recurrent bacterial infections.
4. Asthmatics between the ages of 19 and 80, without a history of recurrent bacterial infections.
5. individuals between the age of 19 and 80 who have a history of frequent bacterial infections and are being evaluated for humoral immunodeficiency.

Exclusion Criteria:

The following groups will be excluded:

1. Subjects who are currently receiving or have ever received immunoglobulin replacement therapy.
2. subjects who are on immune suppressive agents.
3. Subjects who are on chronic steroids or have received an intramuscular injection of steroids in the three months prior to enrollment or oral/intravenous steroids within a month of enrollment or two or more prednisone bursts in the past year.
4. subjects on antiepileptic agents.
5. Subjects who have received the pneumococcal polysaccharide vaccine, PPV-23 6) Pregnant women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from pre-to post-vaccination antibody titer | day one- day of vaccine and one month later
  Evaluate the immune response in the 5 groups of subjects

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States